CLINICAL TRIAL: NCT02718911
Title: A Phase 1a/1b Trial Investigating the CSF-1R Inhibitor LY3022855 in Combination With Durvalumab (MEDI4736) or Tremelimumab in Patients With Advanced Solid Tumors
Brief Title: A Study of LY3022855 in Combination With Durvalumab or Tremelimumab in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 16348; I5F-MC-JSCC (Other: Eli Lilly and Company); 2016-000427-11 (EudraCT Number)
Record Dates: First submitted 2016-03-21; First posted 2016-03-24 (Estimated); Results first posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Solid Tumor
MeSH Terms: interventions — LY3022855; durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LY3022855 + Durvalumab (Dose Escalation) (Experimental): Cohort D1A: LY3022855 (25 mg,QW)+Durvalumab (750mg,Q2W):
  25 mg LY3022855 administered once weekly (QW) intravenously (IV) in combination with 750 mg durvalumab administered every 2 weeks (Q2W) IV. Treatment may continue until disease progression or discontinuation.
  Cohort D2A: LY3022855 (50 mg,QW)+Durvalumab (750mg,Q2W) 50 mg LY3022855 administered QW intravenously (IV) in combination with 750 mg durvalumab administered Q2W IV. Treatment may continue until disease progression or discontinuation.
  Cohort D3A: LY3022855 (75 mg,QW)+Durvalumab (750mg,Q2W) 75 mg LY3022855 administered QW intravenously (IV) in combination with 750 mg durvalumab administered Q2W IV. Treatment may continue until disease progression or discontinuation.
  Cohort D4A: LY3022855 (100 mg,QW)+Durvalumab (750mg,Q2W) 100 mg LY3022855 administered QW intravenously (IV) in combination with 750 mg durvalumab administered Q2W IV. Treatment may continue until disease progression or discontinuation.
  Interventions: Drug: LY3022855; Drug: Durvalumab
- LY3022855 + Tremelimumab (Dose Escalation) (Experimental): Cohort T1A: LY3022855 (50 mg,QW) +Tremelimumab (75mg,Q4W):
  50 mg LY3022855 administered QW intravenously (IV) in combination with 75 mg tremelimumab administered every 4 weeks (Q4W) IV. Treatment may continue until disease progression or discontinuation.
  Cohort T2A: LY3022855 (100 mg,QW) +Tremelimumab (75mg,Q4W) 100 mg LY3022855 administered QW intravenously (IV) in combination with 75 mg tremelimumab administered Q4W IV. Treatment may continue until disease progression or discontinuation.
  Cohort T3A: LY3022855 (100 mg,QW) +Tremelimumab (225 mg,Q4W) 100 mg LY3022855 administered QW intravenously (IV) in combination with 225 mg tremelimumab administered Q4W IV. Treatment may continue until disease progression or discontinuation.
  Cohort T4A: LY3022855 (100 mg,QW) +Tremelimumab (750 mg,Q4W) 100 mg LY3022855 administered QW intravenously (IV) in combination with 750 mg tremelimumab administered Q4W IV. Treatment may continue until disease progression or discontinuation.
  Interventions: Drug: LY3022855; Drug: Tremelimumab
- LY3022855 + Durvalumab (Expansion) (Experimental): Cohort B-1: NSCLC LY3022855+ Durvalumab:
  100 mg LY3022855 administered QW intravenously (IV) in combination with 750 mg durvalumab administered Q2W IV. Treatment may continue until disease progression or discontinuation.
  Cohort B-1: OVARIAN LY3022855+ Durvalumab:
  100 mg LY3022855 administered QW intravenously (IV) in combination with 750 mg durvalumab administered Q2W IV. Treatment may continue until disease progression or discontinuation.
  Interventions: Drug: LY3022855; Drug: Durvalumab

INTERVENTIONS:
Drug: LY3022855 — Administered IV
Drug: Durvalumab — Administered IV
  Other Names: MEDI4736
  Arms: LY3022855 + Durvalumab (Dose Escalation); LY3022855 + Durvalumab (Expansion)
Drug: Tremelimumab — Administered IV
  Arms: LY3022855 + Tremelimumab (Dose Escalation)

SUMMARY:
The main purpose of this study is to evaluate the safety of the colony-stimulating factor 1 receptor (CSF-1R) inhibitor LY3022855 in combination with durvalumab or tremelimumab in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Must have histological or cytological evidence of a diagnosis of cancer that is not amenable to curative therapy.
* Part B: Must have a type of malignancy that is being studied.
* Part A and Part B (ovarian cancer cohort only): Must be willing to undergo pretreatment and on-treatment core needle or excisional tumor biopsies.
* Part A (all cohorts): Have the presence of measureable and /or nonmeasurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Part B (all cohorts): Have the presence of measurable disease as defined by the RECIST 1.1.
* Have adequate normal organ and marrow function, including the following:

  * Absolute neutrophil count ≥ 1.5 x 10⁹/Liters (L) (1500/cubic millimeters)
  * Platelet count ≥ 100 x 10⁹/L (≥100,000/cubic millimeters)
  * Hemoglobin ≥9 grams per deciliter or ≥5.6 millimoles per liter
  * Serum Creatinine ≤1.5 × institutional upper limit of normal (ULN)
  * Total bilirubin ≤1.5 × institutional ULN
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × institutional ULN OR ≤5 × institutional ULN for participants with liver metastases
  * International normalized ratio (INR) or prothrombin time (PT) INR ≤1.5 × institutional ULN or PT ≤5 seconds above institutional ULN
  * PTT or activated partial thromboplastin time (aPTT) ≤5 seconds above institutional ULN
  * Thyroid stimulating hormone (TSH) OR free thyroxine (T4) within the normal limits
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale.

Exclusion Criteria:

* Are currently receiving or have had prior use of immunosuppressive medication within 28 days before the first dose of study drug, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 milligrams/day of prednisone, or an equivalent corticosteroid.
* Have symptomatic central nervous system (CNS) malignancy or metastasis.
* Have had any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, have any unresolved irAE Grade >1, or any irAE that led to the permanent discontinuation of prior immunotherapy.
* Have experienced a Grade ≥3 AE or a neurologic or ocular AE of any grade while receiving prior immunotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- United States (7):
  - Sarah Cannon Research Institute at HealthOne, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Winship Cancer Center Emory University, Atlanta, Georgia
  - New York University Medical Center, New York, New York
  - Columbia University College of Phys & Surgeons, New York, New York
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - GZA St Augustinus, Wilrijk
- Masarykuv Onkology Institute, Brno, Czech Republic, Czechia
- Israel (3):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Falchook GS, Peeters M, Rottey S, Dirix LY, Obermannova R, Cohen JE, Perets R, Frommer RS, Bauer TM, Wang JS, Carvajal RD, Sabari J, Chapman S, Zhang W, Calderon B, Peterson DA. A phase 1a/1b trial of CSF-1R inhibitor LY3022855 in combination with durvalumab or tremelimumab in patients with advanced solid tumors. Invest New Drugs. 2021 Oct;39(5):1284-1297. doi: 10.1007/s10637-021-01088-4. Epub 2021 Apr 14. PMID 33852104
- See also: Click here for more information about this study: A Study of LY3022855 in Combination With Durvalumab or Tremelimumab in Participants With Advanced Solid Tumors — https://trials.lilly.com/en-US/find/completed?trialname=I5F-MC-JSCC&externalRequestID=68cbce79-fbf1-46c5-852a-338ca6e2be85

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study has two parts:
  Part A: Dose-escalation of LY3022855 combined with durvalumab or tremelimumab.
  Part B: Dose-expansion of LY3022855 combined with durvalumab.
Groups:
- Cohort D1A: LY3022855 (25 mg,QW)+Durvalumab (750mg,Q2W): 25 mg LY3022855 administered once weekly (QW) intravenously (IV) in combination with 750 mg durvalumab administered every 2 weeks (Q2W) IV. Treatment may continue until disease progression or discontinuation.
- Cohort D2A: LY3022855 (50 mg,QW)+Durvalumab (750mg,Q2W): 50 mg LY3022855 administered QW intravenously (IV) in combination with 750 mg durvalumab administered Q2W IV. Treatment may continue until disease progression or discontinuation.
- Cohort D3A: LY3022855 (75 mg,QW)+Durvalumab (750mg,Q2W): 75 mg LY3022855 administered QW intravenously (IV) in combination with 750 mg durvalumab administered Q2W IV. Treatment may continue until disease progression or discontinuation.
- Cohort D4A: LY3022855 (100 mg,QW)+Durvalumab (750mg,Q2W): 100 mg LY3022855 administered QW intravenously (IV) in combination with 750 mg durvalumab administered Q2W IV. Treatment may continue until disease progression or discontinuation.
- Cohort T1A: LY3022855 (50 mg,QW) +Tremelimumab (75mg,Q4W): 50 mg LY3022855 administered QW intravenously (IV) in combination with 75 mg tremelimumab administered every 4 weeks (Q4W) IV. Treatment may continue until disease progression or discontinuation.
- Cohort T2A: LY3022855 (100 mg,QW) +Tremelimumab (75mg,Q4W): 100 mg LY3022855 administered QW intravenously (IV) in combination with 75 mg tremelimumab administered Q4W IV. Treatment may continue until disease progression or discontinuation.
- Cohort T3A: LY3022855 (100 mg,QW) +Tremelimumab (225 mg,Q4W): 100 mg LY3022855 administered QW intravenously (IV) in combination with 225 mg tremelimumab administered Q4W IV. Treatment may continue until disease progression or discontinuation.
- Cohort T4A: LY3022855 (100 mg,QW) +Tremelimumab (750 mg,Q4W): 100 mg LY3022855 administered QW intravenously (IV) in combination with 750 mg tremelimumab administered Q4W IV. Treatment may continue until disease progression or discontinuation.
- Cohort B-1: NSCLC LY3022855+ Durvalumab: Cohort B-1: NSCLC
  100 mg LY3022855 administered QW intravenously (IV) in combination with 750 mg durvalumab administered Q2W IV. Treatment may continue until disease progression or discontinuation.
- Cohort B-1: OVARIAN LY3022855+ Durvalumab: Cohort B-1: OVARIAN
  100 mg LY3022855 administered QW intravenously (IV) in combination with 750 mg durvalumab administered Q2W IV. Treatment may continue until disease progression or discontinuation.
Period: Overall Study
Arm/Group | Cohort D1A: LY3022855 (25 mg,QW)+Durvalumab (750mg,Q2W) | Cohort D2A: LY3022855 (50 mg,QW)+Durvalumab (750mg,Q2W) | Cohort D3A: LY3022855 (75 mg,QW)+Durvalumab (750mg,Q2W) | Cohort D4A: LY3022855 (100 mg,QW)+Durvalumab (750mg,Q2W) | Cohort T1A: LY3022855 (50 mg,QW) +Tremelimumab (75mg,Q4W) | Cohort T2A: LY3022855 (100 mg,QW) +Tremelimumab (75mg,Q4W) | Cohort T3A: LY3022855 (100 mg,QW) +Tremelimumab (225 mg,Q4W) | Cohort T4A: LY3022855 (100 mg,QW) +Tremelimumab (750 mg,Q4W) | Cohort B-1: NSCLC LY3022855+ Durvalumab | Cohort B-1: OVARIAN LY3022855+ Durvalumab
Started | 4 | 3 | 3 | 5 | 3 | 5 | 5 | 5 | 19 | 20
Received at Least One Dose of Study Drug | 4 | 3 | 3 | 5 | 3 | 5 | 5 | 5 | 19 | 20
Completed | 0 | 0 | 0 | 4 | 1 | 2 | 2 | 2 | 7 | 1
Not Completed | 4 | 3 | 3 | 1 | 2 | 3 | 3 | 3 | 12 | 19
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Death | 2 | 3 | 1 | 0 | 1 | 3 | 1 | 1 | 4 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 4
Not completed — Reason Not Collected | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 4 | 9

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Cohort D1A: LY3022855 (25 mg,QW)+Durvalumab (750mg,Q2W): 25 mg LY3022855 administered QW intravenously (IV) in combination with 750 mg durvalumab administered Q2W IV. Treatment may continue until disease progression or discontinuation.
- Cohort T1A: LY3022855 (50 mg,QW) +Tremelimumab (75mg,Q4W): 50 mg LY3022855 administered QW intravenously (IV) in combination with 75 mg tremelimumab administered Q4W IV. Treatment may continue until disease progression or discontinuation.
- Total: Total of all reporting groups
Arm/Group | Cohort D1A: LY3022855 (25 mg,QW)+Durvalumab (750mg,Q2W) | Cohort D2A: LY3022855 (50 mg,QW)+Durvalumab (750mg,Q2W) | Cohort D3A: LY3022855 (75 mg,QW)+Durvalumab (750mg,Q2W) | Cohort D4A: LY3022855 (100 mg,QW)+Durvalumab (750mg,Q2W) | Cohort T1A: LY3022855 (50 mg,QW) +Tremelimumab (75mg,Q4W) | Cohort T2A: LY3022855 (100 mg,QW) +Tremelimumab (75mg,Q4W) | Cohort T3A: LY3022855 (100 mg,QW) +Tremelimumab (225 mg,Q4W) | Cohort T4A: LY3022855 (100 mg,QW) +Tremelimumab (750 mg,Q4W) | Cohort B-1: NSCLC LY3022855+ Durvalumab | Cohort B-1: OVARIAN LY3022855+ Durvalumab | Total
Number analyzed (Participants) | 4 | 3 | 3 | 5 | 3 | 5 | 5 | 5 | 19 | 20 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (5.7) | 68.7 (13.4) | 59.0 (10.8) | 56.8 (6.4) | 59.3 (7.1) | 55.2 (20.1) | 62.4 (11.7) | 60.6 (9.6) | 62.5 (8.5) | 55.8 (15.0) | 59.7 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 3 | 2 | 2 | 3 | 2 | 8 | 20 | 45
  Male | 3 | 2 | 0 | 2 | 1 | 3 | 2 | 3 | 11 | 0 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 4
  Not Hispanic or Latino | 4 | 3 | 3 | 4 | 3 | 4 | 3 | 4 | 19 | 19 | 66
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  White | 4 | 2 | 3 | 4 | 3 | 5 | 3 | 3 | 19 | 20 | 66
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 11 | 19
  Czechia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Israel | 0 | 0 | 0 | 1 | 2 | 3 | 2 | 1 | 5 | 5 | 19
  United States | 4 | 3 | 3 | 4 | 1 | 2 | 3 | 4 | 5 | 4 | 33

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose of LY3022855 Combined With Durvalumab (Maximum Tolerated Dose [MTD])
Description: Recommended Phase 2 dose of LY3022855 that could be safely administered in combination with Durvalumab was based on defined dose limiting toxicities (DLT) assessment and MTD definition. MTD is defined as the highest tested dose that has less than 33% probability of causing a DLT.
Time Frame: Cycle 1 (4 weeks)
Population: All participants who received at least one dose of study drug LY3022855 + Durvalumab.
Measure: Number; unit: milligrams (mg)
Groups:
- LY3022855 + Durvalumab: Cohort D1A: 25 mg LY3022855 administered QW intravenously (IV) in combination with 750 mg durvalumab administered Q2W IV.
  Cohort D2A: 50 mg LY3022855 administered QW intravenously (IV) in combination with 750 mg durvalumab administered Q2W IV.
  Cohort D3A: 75 mg LY3022855 administered QW intravenously (IV) in combination with 750 mg durvalumab administered Q2W IV.
  Cohort D4A: 100 mg LY3022855 administered QW intravenously (IV) in combination with 750 mg durvalumab administered Q2W IV.
  Treatment may continue until disease progression or discontinuation.
Arm/Group | LY3022855 + Durvalumab
Number analyzed (Participants) | 15
milligrams (mg) | 100

2. Secondary Outcome: Percentage of Participants Who Exhibit Complete Response (CR) or Partial Response (PR) [Overall Response Rate (ORR)]
Description: ORR was estimated as the percentage of participants with best response of Complete Response (CR) or Partial Response (PR), based on RECIST version 1.1 divided by the total number of participants. CR is defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. Progressive disease (PD) is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Baseline through Measured Progressive Disease or Death (Up To 24 months)
Population: All participants who received at least one dose of study drug.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort D1A: LY3022855 (25 mg,QW)+Durvalumab (750mg,Q2W) | Cohort D2A: LY3022855 (50 mg,QW)+Durvalumab (750mg,Q2W) | Cohort D3A: LY3022855 (75 mg,QW)+Durvalumab (750mg,Q2W) | Cohort D4A: LY3022855 (100 mg,QW)+Durvalumab (750mg,Q2W) | Cohort T1A: LY3022855 (50 mg,QW) +Tremelimumab (75mg,Q4W) | Cohort T2A: LY3022855 (100 mg,QW) +Tremelimumab (75mg,Q4W) | Cohort T3A: LY3022855 (100 mg,QW) +Tremelimumab (225 mg,Q4W) | Cohort T4A: LY3022855 (100 mg,QW) +Tremelimumab (750 mg,Q4W) | Cohort B-1: NSCLC LY3022855+ Durvalumab | Cohort B-1: OVARIAN LY3022855+ Durvalumab
Number analyzed (Participants) | 4 | 3 | 3 | 5 | 3 | 5 | 5 | 5 | 19 | 20
Percentage of participants | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 40.0 [7.6 to 81.1] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 5.0 [0.3 to 21.6]

3. Secondary Outcome: Percentage of Participants Who Exhibit Stable Disease (SD) or CR or PR [Disease Control Rate (DCR)]
Description: DCR is the percentage of participants with a best overall response of CR, PR or SD as defined by RECIST v1.1. CR is defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) for target lesions, no progression of non-target lesions, and no appearance of new lesions. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Baseline through Measured Progressive Disease (Up To 24 months)
Population: All participants who received at least one dose of study drug.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort D1A: LY3022855 (25 mg,QW)+Durvalumab (750mg,Q2W) | Cohort D2A: LY3022855 (50 mg,QW)+Durvalumab (750mg,Q2W) | Cohort D3A: LY3022855 (75 mg,QW)+Durvalumab (750mg,Q2W) | Cohort D4A: LY3022855 (100 mg,QW)+Durvalumab (750mg,Q2W) | Cohort T1A: LY3022855 (50 mg,QW) +Tremelimumab (75mg,Q4W) | Cohort T2A: LY3022855 (100 mg,QW) +Tremelimumab (75mg,Q4W) | Cohort T3A: LY3022855 (100 mg,QW) +Tremelimumab (225 mg,Q4W) | Cohort T4A: LY3022855 (100 mg,QW) +Tremelimumab (750 mg,Q4W) | Cohort B-1: NSCLC LY3022855+ Durvalumab | Cohort B-1: OVARIAN LY3022855+ Durvalumab
Number analyzed (Participants) | 4 | 3 | 3 | 5 | 3 | 5 | 5 | 5 | 19 | 20
Percentage of participants | 75.0 [24.9 to 98.7] | 33.3 [1.7 to 86.5] | 66.7 [13.5 to 98.3] | 80.0 [34.3 to 99.0] | 33.3 [1.7 to 86.5] | 20.0 [1.0 to 65.7] | 20.0 [1.0 to 65.7] | 40.0 [7.6 to 81.1] | 21.1 [7.5 to 41.9] | 25.0 [10.4 to 45.6]

4. Secondary Outcome: Number of Participants With Anti-LY3022855, Anti-Durvalumab or Anti-Tremelimumab Antibodies
Description: Number of participants with positive Anti-LY3022855, Anti-Durvalumab or Anti-Tremelimumab Antibodies was summarized by cohorts.
Time Frame: Baseline through Follow-up (Up To 24 Months)
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D1A: LY3022855 (25 mg,QW)+Durvalumab (750mg,Q2W) | Cohort D2A: LY3022855 (50 mg,QW)+Durvalumab (750mg,Q2W) | Cohort D3A: LY3022855 (75 mg,QW)+Durvalumab (750mg,Q2W) | Cohort D4A: LY3022855 (100 mg,QW)+Durvalumab (750mg,Q2W) | Cohort T1A: LY3022855 (50 mg,QW) +Tremelimumab (75mg,Q4W) | Cohort T2A: LY3022855 (100 mg,QW) +Tremelimumab (75mg,Q4W) | Cohort T3A: LY3022855 (100 mg,QW) +Tremelimumab (225 mg,Q4W) | Cohort T4A: LY3022855 (100 mg,QW) +Tremelimumab (750 mg,Q4W) | Cohort B-1: NSCLC LY3022855+ Durvalumab | Cohort B-1: OVARIAN LY3022855+ Durvalumab
Number analyzed (Participants) | 4 | 3 | 3 | 5 | 3 | 5 | 5 | 5 | 19 | 20
Participants | 0 | 0 | 1 | 1 | 1 | 2 | 3 | 2 | 1 | 7

5. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3022855 in Combination With Either Durvalumab or Tremelimumab, and the Single-Dose
Description: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3022855 in Combination with either Durvalumab or Tremelimumab, and the Single-Dose
Time Frame: Cycle 1 Day 1: 2 hours post End of Infusion (EOI), Day 2: 24-hour post EOI, Day 3: 48 hour post EOI; Cycle 2 Day 8: 2 h post-EOI, Day 9: 24 h post-EOI, Day 10: 48 h post-EOI
Population: All participants who received at least one dose of study drug and had evaluable PK data. Cohort B-1 NSCLC and Cohort B-1 OVARIAN data were combined because they are escalating cohort and the participants are received the same dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (ug/mL)
Groups:
- All LY3022855 (100 mg,QW)+Durvalumab (750mg,Q2W): 100 mg LY3022855 administered QW intravenously (IV) in combination with 750 mg durvalumab administered Q2W IV.
  Cohort B-1 NSCLC:
  100 mg LY3022855 administered QW intravenously (IV) in combination with 750 mg durvalumab administered Q2W IV.
  Cohort B-1 OVARIAN:
  100 mg LY3022855 administered QW intravenously (IV) in combination with 750 mg durvalumab administered Q2W IV. Treatment may continue until disease progression or discontinuation.
Arm/Group | Cohort D1A: LY3022855 (25 mg,QW)+Durvalumab (750mg,Q2W) | Cohort D2A: LY3022855 (50 mg,QW)+Durvalumab (750mg,Q2W) | Cohort D3A: LY3022855 (75 mg,QW)+Durvalumab (750mg,Q2W) | All LY3022855 (100 mg,QW)+Durvalumab (750mg,Q2W) | Cohort T1A: LY3022855 (50 mg,QW) +Tremelimumab (75mg,Q4W) | Cohort T2A: LY3022855 (100 mg,QW) +Tremelimumab (75mg,Q4W) | Cohort T3A: LY3022855 (100 mg,QW) +Tremelimumab (225 mg,Q4W) | Cohort T4A: LY3022855 (100 mg,QW) +Tremelimumab (750 mg,Q4W)
Number analyzed (Participants) | 4 | 3 | 3 | 44 | 3 | 5 | 5 | 5
micrograms per milliliter (ug/mL)
  Cycle 1 | 5.33 (46) | 11.9 (72) | 23.8 (22) | 32.9 (28) | 13.8 (30) | 32 (30) | 30.3 (25) | 27 (34)
  Cycle 2:: number analyzed (Participants) | 3 | 3 | 3 | 29 | 3 | 3 | 0 | 3
  Cycle 2: | 5.11 (61) | 16.6 (8) | 35.3 (17) | 43.1 (38) | 15.1 (33) | 44.4 (39) |  | 30.7 (16)

ADVERSE EVENTS:
Time Frame: Up To 30 Months
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At risk adjusted accordingly.
Arm/Group | Cohort D1A: LY3022855 (25 mg,QW)+Durvalumab (750mg,Q2W) | Cohort D2A: LY3022855 (50 mg,QW)+Durvalumab (750mg,Q2W) | Cohort D3A: LY3022855 (75 mg,QW)+Durvalumab (750mg,Q2W) | Cohort D4A: LY3022855 (100 mg,QW)+Durvalumab (750mg,Q2W) | Cohort T1A: LY3022855 (50 mg,QW) +Tremelimumab (75mg,Q4W) | Cohort T2A: LY3022855 (100 mg,QW) +Tremelimumab (75mg,Q4W) | Cohort T3A: LY3022855 (100 mg,QW) +Tremelimumab (225 mg,Q4W) | Cohort T4A: LY3022855 (100 mg,QW) +Tremelimumab (750 mg,Q4W) | Cohort B-1: NSCLC LY3022855+ Durvalumab | Cohort B-1: OVARIAN LY3022855+ Durvalumab
All-Cause Mortality (participants affected / at risk) | 2/4 | 3/3 | 1/3 | 0/5 | 1/3 | 3/5 | 1/5 | 1/5 | 4/19 | 3/20
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/3 | 1/5 | 0/3 | 2/5 | 3/5 | 3/5 | 12/19 | 5/20
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 5/5 | 3/3 | 5/5 | 5/5 | 5/5 | 19/19 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort D1A: LY3022855 (25 mg,QW)+Durvalumab (750mg,Q2W) (N=4) | Cohort D2A: LY3022855 (50 mg,QW)+Durvalumab (750mg,Q2W) (N=3) | Cohort D3A: LY3022855 (75 mg,QW)+Durvalumab (750mg,Q2W) (N=3) | Cohort D4A: LY3022855 (100 mg,QW)+Durvalumab (750mg,Q2W) (N=5) | Cohort T1A: LY3022855 (50 mg,QW) +Tremelimumab (75mg,Q4W) (N=3) | Cohort T2A: LY3022855 (100 mg,QW) +Tremelimumab (75mg,Q4W) (N=5) | Cohort T3A: LY3022855 (100 mg,QW) +Tremelimumab (225 mg,Q4W) (N=5) | Cohort T4A: LY3022855 (100 mg,QW) +Tremelimumab (750 mg,Q4W) (N=5) | Cohort B-1: NSCLC LY3022855+ Durvalumab (N=19) | Cohort B-1: OVARIAN LY3022855+ Durvalumab (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort D1A: LY3022855 (25 mg,QW)+Durvalumab (750mg,Q2W) (N=4) | Cohort D2A: LY3022855 (50 mg,QW)+Durvalumab (750mg,Q2W) (N=3) | Cohort D3A: LY3022855 (75 mg,QW)+Durvalumab (750mg,Q2W) (N=3) | Cohort D4A: LY3022855 (100 mg,QW)+Durvalumab (750mg,Q2W) (N=5) | Cohort T1A: LY3022855 (50 mg,QW) +Tremelimumab (75mg,Q4W) (N=3) | Cohort T2A: LY3022855 (100 mg,QW) +Tremelimumab (75mg,Q4W) (N=5) | Cohort T3A: LY3022855 (100 mg,QW) +Tremelimumab (225 mg,Q4W) (N=5) | Cohort T4A: LY3022855 (100 mg,QW) +Tremelimumab (750 mg,Q4W) (N=5) | Cohort B-1: NSCLC LY3022855+ Durvalumab (N=19) | Cohort B-1: OVARIAN LY3022855+ Durvalumab (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 6 (16) | 6 (14)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Atrial enlargement (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac discomfort (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Meibomianitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 6 (8)
Swelling of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (5)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 2 (4) | 2 (2) | 2 (3) | 4 (4)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 3 (4)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (3) | 2 (4) | 1 (1) | 3 (5) | 5 (7) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lip blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (6) | 7 (12) | 9 (15)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (6) | 4 (8)
Administration site coldness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Catheter site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site scab (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Early satiety (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (6) | 5 (5)
Fatigue (General disorders) | 3 (4) | 3 (5) | 3 (4) | 3 (3) | 1 (1) | 2 (2) | 3 (5) | 2 (3) | 8 (11) | 11 (18)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nodule (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 3 (6) | 5 (6)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 4 (6) | 4 (5)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (6) | 0 (0) | 2 (2) | 4 (5) | 7 (14)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 2 (6) | 4 (6)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 1 (1) | 1 (2) | 1 (3) | 2 (3) | 7 (13) | 10 (30)
Aspiration pleural cavity (Investigations) | 1 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (3) | 4 (7) | 1 (2)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (4) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 2 (6) | 3 (22) | 0 (0) | 3 (18) | 2 (6) | 3 (7) | 6 (15) | 9 (22)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (6) | 2 (6)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram repolarisation abnormality (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (4)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (4) | 3 (5)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Qrs axis abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 3 (5) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 10 (11) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 2 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 2 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (12) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 1 (1) | 1 (6) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 4 (9) | 1 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (5)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 3 (3)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 3 (5)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drooling (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 5 (13)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coital bleeding (Reproductive system and breast disorders) | 1/1 (1) | 0/1 (0) | 0 (0) | 0/3 (0) | 0/2 (0) | 0/2 (0) | 0/3 (0) | 0/2 (0) | 0/8 (0) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 2 (2) | 2 (4) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 4 (6)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Pulmonary venous thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hair growth rate abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (6) | 3 (3) | 3 (9) | 1 (4) | 1 (1) | 3 (5) | 1 (8) | 2 (2) | 3 (6)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (5)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 1 (11) | 2 (3) | 1 (1) | 2 (2) | 3 (6) | 2 (5) | 1 (3) | 3 (9)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (10) | 7 (9)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT02718911/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-21): https://cdn.clinicaltrials.gov/large-docs/11/NCT02718911/SAP_001.pdf